CLINICAL TRIAL: NCT04182100
Title: Phase 2 Single Arm Study of Efficacy and Safety of P1101 for Polycythemia Vera (PV) Patients for Whom the Current Standard of Treatment is Difficult to Apply
Brief Title: Efficacy and Safety of P1101 in Polycythemia Vera Patients for Whom the Standard of Treatment is Difficult to Apply
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PharmaEssentia Japan K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A19-201
Record Dates: First submitted 2019-11-15; First posted 2019-12-02 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2021-12

CONDITIONS: Polycythemia Vera (PV)
Keywords: Myeloproliferative Neoplasms
MeSH Terms: conditions — Polycythemia Vera; Myeloproliferative Disorders | interventions — Aspirin; Phlebotomy

STUDY DESIGN:
Intervention Model Description: Conventional treatment based on phlebotomies, low-dose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of P1101 (ropeginterferon alfa-2b) once every 2 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- P1101 (Experimental): Conventional treatment based on phlebotomies, low-dose aspirin (acetylsalicylic acid, 75-150 mg/day) plus the subcutaneous administration of pegylated proline-interferon alpha-2b (P1101, ropeginterferon alfa-2b) once every 2 weeks.
  Interventions: Drug: P1101; Drug: Low-dose aspirin; Procedure: Phlebotomy

INTERVENTIONS:
Drug: P1101 — P1101 (ropeginterferon alfa-2b) will be administered subcutaneously every 2 weeks at the starting dose of 100 μg every two weeks (or 50 μg in patients under another cytoreductive therapy). The dose should be gradually increased by 50 μg every two weeks (in parallel, other cytoreductive therapy should be decreased gradually, as appropriate) until stabilization of the hematological parameters is achieved (hematocrit <45%, platelets <400 x 10^9/L and leukocytes <10 x 10^9/L). The maximum recommended single dose is 500 μg injected every two weeks. The dose will be maintained at the highest level which can be tolerated and delivers best possible disease response.
  Other Names: ropeginterferon alfa-2b
Drug: Low-dose aspirin — Low-dose aspirin (acetylsalicylic acid) (75-150 mg/day) will be given as background therapy during the 12 months of study treatment, unless contraindicated.
  Other Names: Low-dose acetylsalicylic acid
Procedure: Phlebotomy — Phlebotomy is performed aiming at a hematocrit < 45%. When the hematocrit value is 45% or higher, phlebotomy is performed. The volume of phlebotomy per procedure should be 200 to 400 mL while monitoring the circulatory dynamics such as blood pressure and pulse. In the elderly and patients with cardiovascular disorders, a small volume (100-200 mL) should be considered to avoid rapid changes in hemodynamics.

SUMMARY:
This is a Phase 2 single arm study to investigate efficacy and safety of P1101 for adult Japanese patients with PV.

DETAILED DESCRIPTION:
Eligible patients will be treated with P1101, starting at 100 μg (or 50 μg in patients under another cytoreductive therapy). The dose should be gradually increased by 50 μg every two weeks (in parallel, other cytoreductive therapy should be decreased gradually, as appropriate) until stabilization of the hematological parameters is achieved (hematocrit <45%, platelets <400 x 10^9/L and leukocytes <10 x 10^9/L). The maximum recommended single dose is 500 μg injected every two weeks.

At week 36 (month 9) and week 52 (month 12), the primary study endpoint, phlebotomy-free CHR, will be analyzed. After completion of the 52-week study duration, provision and administration of P1101, collection of the long-term follow up information (blood parameters, molecular and cytogenetic data, safety parameters and as also the optional bone marrow data) will be continued until the drug becomes commercially available for all study subjects..

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥20 years old
2. Patients diagnosed with PV according to the WHO 2008 or WHO 2016 criteria
3. PV patients for whom the current standard of treatment is difficult to apply. (Patients with a documented history of refractory to HU are excluded.)

   * Younger patients (long-term treatment is anticipated)
   * Patients who are categorized as low risk, but cytoreduction is recommended due to disease-related signs and symptoms (headache, dizziness, pruritus, night sweats, fatigue, erythromelalgia, vision disorders, scintillating scotoma, early satiety, abdominal distension).
   * Patients with HU intolerance
4. Total HU treatment duration shorter than 3 years (cumulatively) at screening
5. For cytoreduction naïve patients only: PV in need of cytoreductive treatment, defined by fulfilling as one or more of the following criteria at baseline:

   * at least one previous well documented major cardiovascular PV-related event in the medical history
   * poor tolerance of phlebotomy (defined as a phlebotomy/ procedure-related adverse event causing significant adverse impact on the patient and limiting ability to apply phlebotomy with the intention to keep Hct <45%)
   * frequent need of phlebotomy (more than one phlebotomy within last month prior entering the study)
   * platelet counts greater than 1000 x 10^9/L (for two measurements within the month prior treatment start)
   * leukocytosis (WBC>10 x 10^9/L for two measurements within the month prior treatment start)
6. Adequate hepatic function defined as bilirubin ≤1.5 x upper limit normal (ULN), international normalized ratio (INR) ≤1.5 x ULN, albumin >3.5 g/dL, alanine aminotransferase (ALT) ≤2.0 x ULN, aspartate aminotransferase (AST) ≤2.0 x ULN at screening
7. Hemoglobin (HGB) ≥10 g/dL at screening
8. Neutrophil count ≥1.5 x 10^9/L at screening
9. Serum creatinine ≤1.5 x ULN at screening
10. Hospital Anxiety and Depression Scale (HADS) score 0-7 on both subscales (Patients with a borderline of HADS score [score 7 but <10] or patients with necessity [expected benefits are higher than the risks] based on investigators' discretion are required to receive following assessment by psychiatric specialist to confirm the eligibility for IFNα therapy.).
11. Males and females of childbearing potential, as well as all women <2 years after the onset of menopause, must agree to use an acceptable form of birth control until 28 days following the last dose of the study drug
12. Written informed consent obtained from the patient or the patient's legal representative, and ability for the patient to comply with the requirements of the study

Exclusion Criteria:

1. Patients with symptomatic splenomegaly
2. Previous use of IFNα for any indication
3. Any contraindications or hypersensitivity to interferon-alfa
4. Co-morbidity with severe or serious conditions which may impact patient participation in the study in investigator's opinion
5. History of major organ transplantation
6. Pregnant or lactating females
7. Patients with any other medical conditions, which in the opinion of the Investigator would compromise the results of the study or may impair compliance with the requirements of the protocol

   7-1. History or presence of thyroid dysfunction (clinical symptoms of hyper- or hypo-thyroidism) of the autoimmune origin, except late stages cases on the oral thyroid substitution therapy, where potential exacerbation under interferon therapy will not constitute any further harm to the patient

   7-2.Documented autoimmune disease (e.g., hepatitis, idiopathic thrombocytopenic purpura [ITP], scleroderma, psoriasis, or any autoimmune arthritis)

   7-3. Clinically relevant pulmonary infiltrates and pneumonitis at screening, patients with a history of interstitial pulmonary disease

   7-4. Active infections with systemic manifestations (e.g., bacterial, fungal, hepatitis B [HBV], hepatitis C [HCV], or human immunodeficiency virus [HIV]) at screening)

   7-5. Evidence of severe retinopathy (e.g., cytomegalovirus retinitis [CMV], macular degeneration) or clinically relevant ophthalmological disorder (due to diabetes mellitus or hypertension) based on the ophthalmological assessment by specialists.

   7-6. Uncontrolled depression

   7-7. Previous suicide attempts or at any risk of suicide at screening
8. Uncontrolled diabetes mellitus (HbA1c level of > 7% at baseline)
9. History of any malignancy within for the past 5 years
10. History of alcohol or drug abuse within the last year
11. History or evidence of post polycythemia vera-myelofibrosis (PPV-MF), essential thrombocythemia, or any non-PV MPN
12. Presence of circulating blasts in the peripheral blood within the last 3 months
13. Use of any investigational drug(s), or investigational drug combinations <4 weeks prior to the first dose of study drug or not recovered from effects of prior administration of any investigational agent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2021-03-08 (Actual); Study Completion 2021-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Ehime University Hospital, Toon-shi, Ehime
  - Mie University Hospital, Tsu, Mie-ken
  - Osaka University Hospital, Suita-shi, Osaka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - NTT Medical Center Tokyo, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi

REFERENCES:
- [Derived] Qin A, Shimoda K, Suo S, Fu R, Kirito K, Wu D, Liao J, Chen H, Wu L, Su X, Gao Y, Sato T, Li Y, Zhang J, Shen W, Wang W, Zhang L, Jin J, Komatsu N. Population Pharmacokinetics-Pharmacodynamics and Exposure-Response of Ropeginterferon Alfa-2b in Chinese and Japanese Patients With Polycythemia Vera. Pharmacol Res Perspect. 2025 Jun;13(3):e70109. doi: 10.1002/prp2.70109. PMID 40313042

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was initiated at 8 sites in 1 country.
Pre-assignment Details: Eligible patients were to be treated with P1101, starting at 100 μg (or 50 μg in patients under another cytoreductive therapy). The dose was to be gradually increased by 50 μg every 2 weeks (in parallel, other cytoreductive therapy should be decreased gradually, as appropriate) until stabilization of the hematological parameters is achieved (hematocrit <45%, platelet count ≤400 × 10^9/L, and leukocyte count ≤10 × 10^9/L). The maximum recommended single dose is 500 μg injected every 2 weeks.
Groups:
- P1101: Eligible patients were to be treated with P1101, starting at 100 μg (or 50 μg in patients under another cytoreductive therapy). The dose was to be gradually increased by 50 μg every 2 weeks (in parallel, other cytoreductive therapy should be decreased gradually, as appropriate) until stabilization of the hematological parameters is achieved (hematocrit <45%, platelet count ≤400 × 10^9/L, and leukocyte count ≤10 × 10^9/L). The maximum recommended single dose is 500 μg injected every 2 weeks.At Week 36 (Month 9) and Week 52 (Month 12), the primary study endpoint, phlebotomy-free CHR, was to be analyzed. After completion of the 52-week study period, provision and administration of P1101, collection of the long-term follow up information (blood parameters, molecular and cytogenetic data, safety parameters, and as also the optional bone marrow data) would be continued.
Period: Overall Study
Arm/Group | P1101
Started | 29
Completed | 27
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- P1101: The dose was to be gradually increased by 50 μg every 2 weeks (in parallel, other cytoreductive therapy should be decreased gradually, as appropriate) until stabilization of the hematological parameters is achieved (hematocrit <45%, platelet count ≤400 × 10^9/L, and leukocyte count ≤10 × 10^9/L). The maximum recommended single dose is 500 μg injected every 2 weeks.
Arm/Group | P1101
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Japan | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Who Achieved Durable Phlebotomy-free Complete Hematological Response (CHR) at Month 12
Description: The primary efficacy endpoint was the phlebotomy-free CHR rate at Months 9 and 12.
  The phlebotomy-free CHR rate was defined as the proportion of patients who achieved phlebotomy-free CHR at both Months 9 and 12 without phlebotomies during the previous 3 months.
  A responder in sense of the primary endpoint was a patient who met all of the following criteria at Months 9 and 12:
  Hematocrit <45% phlebotomy-free (absence of phlebotomy during the previous 3 months) Platelet count ≤400 × 10^9/L Leukocyte count ≤10 × 10^9/L
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | P1101
Number analyzed (Participants) | 29
Participants | 8

2. Secondary Outcome: Changes in Hct From Baseline
Description: Hct will be recorded every 3 months.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: Intent-to-Treat (ITT) Population Number analyzed: the number of subjects with non-missing value at the visit
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | P1101
Number analyzed (Participants) | 29
percent
  Baseline | 46.85 (4.369)
  Change from Baseline at Week 12 | -2.21 (4.249)
  Change from Baseline at Week 24: number analyzed (Participants) | 27
  Change from Baseline at Week 24 | -2.95 (6.660)
  Change from Baseline at Week 36: number analyzed (Participants) | 27
  Change from Baseline at Week 36 | -3.09 (5.888)
  Change from Baseline at Week 52: number analyzed (Participants) | 27
  Change from Baseline at Week 52 | -5.45 (6.656)

3. Secondary Outcome: Changes in WBC Count From Baseline
Description: WBC count will be recorded every 3 months.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: Intent-to-Treat (ITT) Population Number analyzed: the number of subjects with non-missing value at the visit
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | P1101
Number analyzed (Participants) | 29
10^9 cells/L
  Baseline | 17.07 (8.824)
  Change from Baseline at Week 12 | -8.50 (7.607)
  Change from Baseline at Week 24: number analyzed (Participants) | 27
  Change from Baseline at Week 24 | -10.57 (7.842)
  Change from Baseline at Week 36: number analyzed (Participants) | 27
  Change from Baseline at Week 36 | -11.29 (8.214)
  Change from Baseline at Week 52: number analyzed (Participants) | 27
  Change from Baseline at Week 52 | -11.71 (8.379)

4. Secondary Outcome: Changes in Plt Count From Baseline
Description: Plt count will be recorded every 3 months.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: Intent-to-Treat (ITT) Population Number analyzed: the number of subjects with non-missing value at the visit
Measure: Mean (Standard Deviation); unit: 10^9 platelets/L
Arm/Group | P1101
Number analyzed (Participants) | 29
10^9 platelets/L
  Baseline | 747.3 (378.32)
  Change from Baseline at Week 12 | -283.6 (325.58)
  Change from Baseline at Week 24: number analyzed (Participants) | 27
  Change from Baseline at Week 24 | -423.0 (377.93)
  Change from Baseline at Week 36: number analyzed (Participants) | 27
  Change from Baseline at Week 36 | -467.4 (396.44)
  Change from Baseline at Week 52: number analyzed (Participants) | 27
  Change from Baseline at Week 52 | -493.6 (374.90)

5. Secondary Outcome: Changes in Spleen Size From Baseline
Description: Spleen size will be recorded every 3 months.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: Intent-to-Treat (ITT) Population Number analyzed: the number of subjects with non-missing value at the visit
Measure: Mean (Standard Deviation); unit: square centimeter
Arm/Group | P1101
Number analyzed (Participants) | 29
square centimeter
  Change from Baseline at Week 12 | 2.587 (9.5810)
  Change from Baseline at Week 24: number analyzed (Participants) | 27
  Change from Baseline at Week 24 | 1.847 (10.8476)
  Change from Baseline at Week 36: number analyzed (Participants) | 27
  Change from Baseline at Week 36 | 2.604 (12.1256)
  Change from Baseline at Week 52: number analyzed (Participants) | 27
  Change from Baseline at Week 52 | 5.043 (15.1477)

6. Secondary Outcome: Time to Requiring no Phlebotomy
Description: Time to requiring no phlebotomy is recorded.
Time Frame: Up to 12 months
Measure: Mean (Inter-Quartile Range); unit: month
Arm/Group | P1101
Number analyzed (Participants) | 29
month
  Baseline | 0.3 [0 to 1]
  Week 12 | 0.1 [0 to 1]
  Week 24 | 0.0 [0 to 1]
  Week 36 | 0.0 [0 to 1]
  Week 52 | 0.0 [0 to 1]

7. Secondary Outcome: Time Required to First Response
Description: Time required to first response is defined as time to achieve complete hematological response (CHR) without phlebotomy.
Time Frame: Up to 12 months
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | P1101
Number analyzed (Participants) | 29
month | 11.90 [5.50 to 12.00]

8. Secondary Outcome: Duration of Response Maintenance
Description: Duration of maintained complete hematologic response (CHR) since first achievement of CHR after administration of the study drug will be calculated.
Time Frame: Up to 12 months
Measure: Mean (Standard Deviation); unit: month
Arm/Group | P1101
Number analyzed (Participants) | 29
month
  Initial response | 3.38 (2.715)
  Longest response | 3.77 (2.881)

9. Secondary Outcome: Proportion of Subjects Without Thrombotic or Hemorrhagic Events
Description: Thrombotic or hemorrhagic events will be recorded any time during the study. The proportion of subjects without thrombotic or hemorrhagic events is defined as the proportion of subjects experienced no thrombotic and hemorrhagic events during the study period (12 months).
Time Frame: Up to 12 months
Population: No thrombotic or hemorrhagic events related to PV were observed throughout the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | P1101
Number analyzed (Participants) | 29
Participants | 0

10. Secondary Outcome: Change of JAK2 Mutant Allelic Burden Over Time vs. Baseline
Description: Quantitative JAK2 measurements at screening, Months 3, 6, 9 and 12 (central laboratory) for subjects who signed consent form. Change of JAK2 allelic burden over time will be assessed.
Time Frame: Baseline, 3 months, 6 months, 9 months and 12 months
Population: Quantitative JAK2 measurements at screening, Months 3, 6, 9 and 12 (central laboratory) for subjects who signed consent form. Change of JAK2 allelic burden over time will be assessed.
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | P1101
Number analyzed (Participants) | 29
percent
  Baseline | 72.1881 (23.30272)
  Change from baseline at Week 12 | -4.9006 (10.14497)
  Change from baseline at Week 24 | -7.4963 (15.72194)
  Change from baseline at Week 36 | -12.4549 (16.32228)
  Change from baseline at Week 52 | -19.1748 (22.64181)

11. Secondary Outcome: PK of P1101
Description: Trough concentration is the measured concentration of a drug at the end of a dosing interval at steady state every 2 weeks.
  Additionally, serum concentration is measured at hours 0, 24, 48, 96 and 168 after administration at Week 0 and Week 28.
Time Frame: Up to 12 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | P1101
Number analyzed (Participants) | 29
ng/mL | 50.3 (17.8)

12. Other Pre Specified Outcome: Status of Bone Marrow Histological Remission (Optional)
Description: Status of bone marrow histological remission defined as the disappearance of hypercellularity (age-adjusted), trilineage growth (panmyelosis) and absence of >grade 1 reticulin fibrosis
Time Frame: 0 month, 12 months
Population: In myelographic findings, Patient 001-006 showed improvement with the disappearance of findings considered to be MPN; Patients 001-009 and 006-002 showed no change in pathological findings; and Patient 001-005 showed evidence of fibrosis.
Measure: Count of Participants; unit: Participants
Arm/Group | P1101
Number analyzed (Participants) | 29
Participants
  Showed no change in pathological findings | 2
  Showed improvement with the disappearance of findings considered to be MPN | 1
  Showed evidence of fibrosis | 1

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: All AEs reported on or after the date of first dose until 30 days (inclusive) after the last dose of the study drug were to be considered treatment-emergent adverse events (TEAEs) and were to be summarized.
Arm/Group | P1101
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 29/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | P1101 (N=29)
Alopecia (Skin and subcutaneous tissue disorders) | 16
Eczema (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 2
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 8
Influenza like illness (General disorders) | 8
Injection site reaction (General disorders) | 4
Pyrexia (General disorders) | 4
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 9
Dental caries (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Chronic gastritis (Gastrointestinal disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Food poisoning (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Hyperaesthesia teeth (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 5
Gastroenteritis (Infections and infestations) | 4
Hordeolum (Infections and infestations) | 2
Appendicitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Dermatophytosis of nail (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dry eye (Eye disorders) | 2
Photophobia (Eye disorders) | 2
Retinal haemorrhage (Eye disorders) | 1
Swelling of eyelid (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Palpitations (Cardiac disorders) | 2
Mitral valve incompetence (Cardiac disorders) | 1
Supraventricular extrasystoles (Cardiac disorders) | 1
Ventricular hypokinesia (Cardiac disorders) | 1
Dizziness (Nervous system disorders) | 2
Headache (Nervous system disorders) | 2
Taste disorder (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Irritability (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Silent thyroiditis (Endocrine disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Chillblains (Injury, poisoning and procedural complications) | 1
Heat illness (Injury, poisoning and procedural complications) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypertonic bladder (Renal and urinary disorders) | 1
Subgaleal haematoma (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04182100/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT04182100/SAP_001.pdf